CLINICAL TRIAL: NCT06855875
Title: Evaluation of Autogenous Tooth- Derived Graft With Bovine Bone For Surgical Repair of Unilateral Alveolar Cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Taha Ibrahim, Ass Prof, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OS-4-23-2
Record Dates: First submitted 2025-02-21; First posted 2025-03-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Cleft
Keywords: teeth derived graft; bovine bone; alveolar cleft grafting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous tooth graft combined with bovine bone (Experimental): This include 8 patients with unilateral alveolar cleft which will be repaired using autogenous tooth graft combined with bovine bone .
  Interventions: Procedure: autogenous tooth graft combined with bovine bone
- bovine bone (Experimental): This include 8 patients in whom alveolar cleft will be repaired using bovine bone .
  Interventions: Procedure: bovine bone

INTERVENTIONS:
Procedure: autogenous tooth graft combined with bovine bone — unilateral alveolar cleft which will be repaired using autogenous tooth graft combined with bovine bone .
  Arms: autogenous tooth graft combined with bovine bone
Procedure: bovine bone — unilateral alveolar cleft which will be repaired using bovine bone .
  Arms: bovine bone

SUMMARY:
The aim of this study is evaluation of autogenous tooth-derived graft combined with bovine bone for surgical repair of unilateral alveolar cleft .

DETAILED DESCRIPTION:
Decalcified dentin graft is thought to be a good graft material that can substitute existing autogenous bone graft materials. It can be easily and readily available, with minimal risk of infection, minimal donor site morbidity as no vital bone is sacrificed, it can be easily shaped to fit into the bony defect and it can be used as block or in powder forms, the hypothesis is to evaluate the biological and the physical properties of both and autogenous tooth derived graft and bovine bone to increase the quality and density of newly formed bone in alveolar cleft grafting

Criteria of patient selection:

Inclusion Criteria:

Patients with unilateral alveolar clefts requiring repair. patients free from any systemic disease that may affect normal healing of bone. patients in an age 7y up to 14 y. patients have teeth to be sacrificed, as primary teeth, carious teeth, malposed teeth, supernumerary tooth& non functional tooth in the study group.

Exclusion criteria:

Bilateral alveolar clefts. Immunocompromized patients. Syndromic patients. Patients have good full set of teeth, cannot be sacrified in study group The patients grouping with unilateral alveolar cleft will be classified into two equal groups according to the grafting material used for alveolar cleft repair.

Study Group:

This will include 8 patients with unilateral alveolar cleft which will be repaired using autogenous tooth graft combined with bovine bone .

Control Group:

This will include 8 patients in whom alveolar cleft will be repaired using bovine bone .

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral alveolar clefts requiring repair.
* patients free from any systemic disease that may affect normal healing of bone.
* patients in an age 7y up to 14 y.
* patients have teeth to be sacrificed, as primary teeth, carious teeth, malposed teeth, supernumerary tooth& non functional tooth in the study group.

Exclusion Criteria:

* Bilateral alveolar clefts.
* Immunocompromized patients.
* Syndromic patients.
* Patients have good full set of teeth, cannot be sacrified in study group

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 1 month
  0 representing no pain and 10 representing the highest level of pain
inflammation score scale | 1 month
  0 no inflammation, 1-3 mild inflammation,4-7 moderate inflammation,8-10 severe inflammation

SECONDARY OUTCOMES:
bone mineral density | 6 months
  density of bone to measure (D1,D2,D3,D4) from 150 HU to 1250HU

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Tanta university, Tanta, Egypt